CLINICAL TRIAL: NCT06277323
Title: UCLA Health Patient Cardiology Care Gaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Richard K. Leuchter, MD, Clinical Instructor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Cardio
Record Dates: First submitted 2024-02-01; First posted 2024-02-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Health Maintenance; Cardiology
Keywords: Cardiology

STUDY DESIGN:
Intervention Model Description: Parallel randomized trial at the physician level.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Quarterly performance email (current state, control condition) (No Intervention): Eligible, randomly assigned physicians will receive status quo quarterly emails with their performance report card.
- Arm 2: Monthly report card only (Experimental): Eligible, randomly assigned physicians will receive behaviorally-informed monthly emails (monthly performance report card) intended to elevate their intentions to improve their performance (i.e., getting more of their patients to close care gaps).
  Interventions: Behavioral: Monthly report card intervention
- Arm 3: Storyboard only (Experimental): Eligible, randomly assigned physicians will receive status quo quarterly emails and get a more visible care gap banner in the electronic health record (EHR), intended to promptly remind them of each patient's care gaps at the start of a patient-physician encounter.
  Interventions: Behavioral: Storyboard intervention
- Arm 4: Monthly report card AND Storyboard (Experimental): Eligible, randomly assigned physicians will receive behaviorally-informed monthly emails and get a more visible care gap banner in the electronic health record (EHR) upon patient encounter.
  Interventions: Behavioral: Monthly report card intervention; Behavioral: Storyboard intervention

INTERVENTIONS:
Behavioral: Monthly report card intervention — The investigators will increase the frequency (monthly instead of quarterly) and enhance the content of the performance feedback emails sent to cardiologists (i.e., behaviorally-informed).
  Arms: Arm 2: Monthly report card only; Arm 4: Monthly report card AND Storyboard
Behavioral: Storyboard intervention — The visibility of the care gap banner in the electronic health record (EHR) upon patient encounter will be enhanced.
  Arms: Arm 3: Storyboard only; Arm 4: Monthly report card AND Storyboard

SUMMARY:
This is a prospective randomized clinical trial evaluating how two behaviorally-informed interventions (i.e., monthly report card and storyboard interventions) impact physician behavior, with the goal of closing care gaps in preventive care and disease management.

In particular, the monthly report card intervention seeks to elevate physicians' intentions to close their patients' care gaps, while the storyboard intervention seeks to prompt action by making patients' care gaps salient. The trial investigates the separate and joint impacts of the proposed behaviorally-informed interventions on encouraging physicians to close their patients' care gaps.

DETAILED DESCRIPTION:
Despite the existence of evidence-based clinical guidelines on how to manage the health of patients with cardiovascular disease that have been shown to improve cardiac function and survival, significant gaps in care persist and optimal medical therapy is often under-utilized. For example, guideline-directed medical therapy (GDMT), statin and aspirin therapy, and blood pressure control are cornerstones of effective management of patients with cardiovascular disease or heart failure. However, current dashboard data indicate that within the UCLA Health system, these medical therapies remain under-utilized.

As part of the quality improvement (QI) initiative sponsored by the Division of Cardiology at UCLA Health, this trial will examine the independent and joint impacts on care gap closure of (1) sending monthly behaviorally-informed emails to physicians with personalized feedback on care gap performance and (2) enhancing the visibility of the open care gaps in the electronic health record upon patient encounter.

Eligible physicians (i.e., UCLA Health Cardiologists) will be randomized to one of four conditions based on a 2 (monthly report card intervention: receive vs. no receive) x 2 (storyboard intervention: receive vs not receive) between-subjects design:

* In the no intervention (control) condition, physician participants will receive quarterly emails with their performance report card (status quo).
* In the monthly report card only condition, behaviorally-informed monthly emails will be sent to inform physicians of their performance and elevate physicians' intentions to get more of their patients to close care gaps.
* In the storyboard only condition, the visibility of care gap banners in the electronic health record (EHR) will be enhanced, which will promptly remind physicians of each patient's care gaps at the start of a patient-physician encounter.
* In the monthly report card and storyboard condition, physicians will receive behaviorally-informed monthly emails and be reminded of each patient's care gaps via the EHR storyboard during patient-physician encounters.

The trial will include physicians participating in an existing UCLA incentive program, as of October 1, 2023, who have a panel size of above 50 patients. In August 2024, new physicians who are eligible for the incentive program and have at least 50 patients in the panel will be randomly assigned into one of the four conditions and become part of the study sample. Randomization will balance for physicians' baseline performance, subspecialty training, years out from training, and estimated panel size.

Monthly performance feedback emails will include physicians' performance on eight cardiology care gaps, their projected earnings in the current quarter and their earnings in the previous quarter. Care gaps include the following: (1) statin or PCSK9 inhibitor use, (2) aspirin use, (3) beta blocker use, (4) angiotensin-converting enzyme inhibitors, angiotensin II receptor blockers, or angiotensin receptor-neprilysin inhibitor use, (5) mineralocorticoid receptor antagonist use, (6) SGLT2i, (7) average HCC/RAF score, and (8) blood pressure control.

Analysis Plan:

* The investigators will use patient-level linear regression models, where the response is a 1/0 indicator of whether the patient has completed any of the open care gaps, with cluster-robust standard errors at the physician level.
* The primary regression model will look at the main effect of the report card intervention and the storyboard intervention.
* In a secondary regression, we will investigate the joint impact of the two interventions, including a report card x storyboard interaction.

Control variables include:

* Patient-level care gap closure (i.e., whether patients closed any of their open care gaps, excluding HCC/RAF score, during the six months before the intervention delivery). For patients who were not in a given physician's panel as of six months before the experiment, mean values across the panel will be imputed.
* Physician characteristics (gender, years out from training, subspecialty training within cardiology) and panel size.
* Patient age (If there will be a missing value, the investigators will replace it with the mean and add a dummy variable to indicate patients with missing age).
* Indicators for patient race/ethnicity (Black non-Hispanic, Hispanic, Asian non-Hispanic, white non-Hispanic, other/mixed, unknown).
* Indicators for patient gender (male, female, other/unknown).
* Indicators for patient 5-digit zip code (all zip codes outside of California will be collapsed into one group).
* Indicators for patient insurance type (Self-pay/uninsured, Medicaid, Medicare Advantage, Medicare Fee For Service, Commercial, VA, Other).

The investigators will conduct subgroup analyses based on:

* Whether the patient is female or male.
* Whether the patient is white non-hispanic or racial/ethnic minority.
* Whether the patient is 65+ (including 65) or below 65 years of age.
* Distance from patient's place of residence to their cardiologist's clinic.
* Whether the patient has commercial or non-commercial insurance.

ELIGIBILITY:
Inclusion criteria:

* Cardiologists who practice at one or more UCLA Health sites in the outpatient setting
* Enrolled in the pre-existing cardiology financial incentive program at UCLA Health
* With patient panel size above 50

Exclusion criteria:

- Cardiologists who were involved in the design of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Care gap closure (patients seen) | 6 months after each patient's first encounter with the physician during the first 12 months of the intervention period
  Whether a patient completed any of the following seven care gaps will be tracked for each patient who visits a physician during the first 12 months of the intervention period: (1) statin or PCSK9 inhibitor use, (2) aspirin use, (3) beta blocker use, (4) angiotensin-converting enzyme inhibitors, angiotensin II receptor blockers, or angiotensin receptor-neprilysin inhibitor use, (5) mineralocorticoid receptor antagonist use, (6) SGLT2i use, and (7) blood pressure control.

SECONDARY OUTCOMES:
Care gap closure (all patients in panel) | 12 months after the intervention starts (for existing patients) or 12 months since patients join the panel (for patients who join during the first six months of the experiment)
  Whether a patient completed any of the following seven care gaps will be tracked for each patient who is in a physician's panel during the first six months of the intervention period: (1) statin or PCSK9 inhibitor use, (2) aspirin use, (3) beta blocker use, (4) angiotensin-converting enzyme inhibitors, angiotensin II receptor blockers, or angiotensin receptor-neprilysin inhibitor use, (5) mineralocorticoid receptor antagonist use, (6) SGLT2i use, and (7) blood pressure control.
Number of care gaps closed (patients seen) | 6 months after each patient's first encounter with the physician during the first 12 months of the intervention period
  The number of care gaps closed will be tracked for each patient who visits a physician during the first 12 months of the intervention period, considering the following seven care gaps: (1) statin or PCSK9 inhibitor use, (2) aspirin use, (3) beta blocker use, (4) angiotensin-converting enzyme inhibitors, angiotensin II receptor blockers, or angiotensin receptor-neprilysin inhibitor use, (5) mineralocorticoid receptor antagonist use, (6) SGLT2i use, and (7) blood pressure control. The investigators will also analyze the number of care gaps closed when excluding care gap (7) blood pressure control.
Number of care gaps closed (all patients in panel) | 12 months after the intervention starts (for existing patients) or 12 months since patients join the panel (for patients who join during the first six months of the experiment)
  The number of care gaps closed will be tracked for each patient who is in a physician's panel during the six months of the intervention period, considering the following seven care gaps: (1) statin or PCSK9 inhibitor use, (2) aspirin use, (3) beta blocker use, (4) angiotensin-converting enzyme inhibitors, angiotensin II receptor blockers, or angiotensin receptor-neprilysin inhibitor use, (5) mineralocorticoid receptor antagonist use, (6) SGLT2i use, and (7) blood pressure control. The investigators will also analyze the proportion of care gaps closed when excluding care gap (7) blood pressure control.
HCC/RAF care gap closure (all patients in panel) | 12 months after the intervention starts (for existing patients) or 12 months since patients join the panel (for patients who join during the first six months of the experiment)
  Whether HCC/RAF coding was completed will be tracked for each patient that is in a physician's panel during the first 12 months of the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Health Department of Medicine, Quality Office, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make any individual participant data available.